CLINICAL TRIAL: NCT03001557
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study With Open-Label Extension Phase of the Efficacy and Safety of Lemborexant in Subjects With Irregular Sleep-Wake Rhythm Disorder and Mild to Moderate Alzheimer's Disease Dementia
Brief Title: Study of Lemborexant for Irregular Sleep-Wake Rhythm Disorder and Mild to Moderate Alzheimer's Disease Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2006-G000-202; 2017-003306-40 (EudraCT Number)
Record Dates: First submitted 2016-11-16; First posted 2016-12-23 (Estimated); Results first posted 2020-01-14 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-04

CONDITIONS: Irregular Sleep-Wake Rhythm Disorder
Keywords: Mild to Moderate Alzheimer's Disease Dementia; sleep; circadian rhythms
MeSH Terms: interventions — lemborexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Lemborexant 2.5 milligrams (mg) (Experimental): Participants will take one lemborexant 2.5 mg tablet and one lemborexant-matched placebo tablet orally each night for 28 consecutive nights immediately (i.e., within 5 minutes) before the time the participant intends to try to sleep.
  Interventions: Drug: Lemborexant 2.5 mg; Drug: Lemborexant-matched placebo
- Lemborexant 5 mg (Experimental): Participants will take one lemborexant 5 mg tablet and one lemborexant-matched placebo tablet orally each night for 28 consecutive nights immediately (i.e., within 5 minutes) before the time the participant intends to try to sleep.
  Interventions: Drug: Lemborexant 5 mg; Drug: Lemborexant-matched placebo
- Lemborexant 10 mg (Experimental): Participants will take one lemborexant 10 mg tablet and one lemborexant-matched placebo tablet orally each night for 28 consecutive nights immediately (i.e., within 5 minutes) before the time the participant intends to try to sleep.
  Interventions: Drug: Lemborexant 10 mg; Drug: Lemborexant-matched placebo
- Lemborexant 15 mg (Experimental): Participants will take one lemborexant 5 mg tablet and one lemborexant 10 mg tablet orally each night for 28 consecutive nights immediately (i.e., within 5 minutes) before the time the participant intends to try to sleep.
  Interventions: Drug: Lemborexant 10 mg; Drug: Lemborexant 15 mg
- Lemborexant-matched placebo (Placebo Comparator): Participants will take two lemborexant-matched placebo tablets orally each night for 28 consecutive nights immediately (i.e., within 5 minutes) before the time the participant intends to try to sleep.
  Interventions: Drug: Lemborexant-matched placebo

INTERVENTIONS:
Drug: Lemborexant 2.5 mg — Lemborexant 2.5 mg tablets
  Arms: Lemborexant 2.5 milligrams (mg)
Drug: Lemborexant 5 mg — Lemborexant 5 mg tablets
  Arms: Lemborexant 5 mg
Drug: Lemborexant 10 mg — Lemborexant 10 mg tablets
  Arms: Lemborexant 10 mg; Lemborexant 15 mg
Drug: Lemborexant 15 mg — Lemborexant 5 mg and 10 mg tablets
  Arms: Lemborexant 15 mg
Drug: Lemborexant-matched placebo — Lemborexant-matched placebo tablets
  Arms: Lemborexant 10 mg; Lemborexant 2.5 milligrams (mg); Lemborexant 5 mg; Lemborexant-matched placebo

SUMMARY:
This study will be conducted to determine the dose response of lemborexant (LEM) on the change from baseline in actigraphy-derived sleep-related parameters, wake-related parameters, and circadian-rhythm related parameters. Following the eligibility screening period, eligible participants will be assigned at random to 1 of 4 doses of LEM or to placebo for 4 weeks. After a 2-week follow-up period, eligible participants may enter an open-label extension period for up to 30 months or until the program discontinuation.

ELIGIBILITY:
Inclusion Criteria (Core Study):

* Male or female, age 60 to 90 years at the time of informed consent
* Able to provide informed consent. If a participant lacks capacity to consent in the investigator's opinion, the participant's assent should be obtained, if required in accordance with local laws, regulations and customs, and the written informed consent of a legal representative should be obtained (capacity to consent and definition of legal representative should be determined in accordance with applicable local laws and regulations).
* Documentation of diagnosis with Alzheimer's disease dementia (AD-D) on the basis of the National Institute on Aging/Alzheimer's Association Diagnostic Guidelines
* Mini Mental State Examination 10 to 26 at Screening
* Meets criteria for Circadian Rhythm Sleep Disorder, Irregular Sleep-Wake Type (Diagnostic and Statistical Manual of Mental Disorders - 5th edition) and the 10th revision of the International Classification of Diseases, as follows: Complaint by the participant or caregiver of difficulty sleeping during the night and/or excessive daytime sleepiness associated with multiple irregular sleep bouts during a 24-hour period
* Frequency of complaint of sleep and wake fragmentation ≥3 days per week
* Duration of complaint of sleep and wake fragmentation ≥3 months
* During the Screening Period, mean actigraphy-derived sleep efficiency (aSE) <87.5% within the defined nocturnal sleep period and mean actigraphy-derived wake efficiency (aWE) <87.5% during the defined wake period
* Confirmation by actigraphy of a combination of sleep bouts of >10 minutes during the wake period plus wake bouts of >10 minutes during the sleep period, totaling at least 4 bouts per 24 hours period, ≥ 3 days per week
* Ambulatory and living in the community or in a residence not classified as a skilled nursing facility (an assisted living facility with separate living quarters where participants and their caregivers reside is acceptable)
* Willing not to start a behavioral or other treatment program for sleep or wake difficulties and not to start a new treatment for other symptoms of AD-D during participation in the study
* Has a reliable and competent caregiver (or caregiver and informants) who can accompany the participant to study visits, administer study medication on a nightly basis and provide information on the status of the participant
* For participants taking a cholinesterase inhibitor and/or memantine, dosing regimen must have been stable for at least 3 months

Inclusion Criteria (Extension Phase):

* Completed the Core Study (End of Study [EOS] Visit). Participants who participated in the Core Study and completed the EOS Visit within 30 days may return to participate in the Extension Phase as long as there are no contraindications due to ongoing adverse events or prohibited medications.

Inclusion Criteria for Caregivers:

* Able to provide informed consent
* Spends at least 10 hours per week with the participant
* Able to meet caregiver requirements
* Willing to provide information on himself/herself regarding sleep quality and caregiver Burden

Exclusion Criteria:

* A diagnosis of vascular dementia, dementia following multiple strokes, or any synucleinopathy / Lewy body disorder. This includes Dementia with Lewy Bodies and Parkinson's disease with or without dementia.
* A current diagnosis of moderate to severe obstructive sleep apnea (OSA) or central sleep apnea, or current use of continuous positive airways pressure even if mild severity of OSA, restless legs syndrome, periodic limb movement disorder (with awakenings), or narcolepsy
* An Apnea-Hypopnea Index or equivalent ≥15 events/hour on diagnostic sleep study conducted prior to Baseline or within 6 months of Screening
* A clinically significant movement disorder that would affect the differentiation of sleep and wake by the actigraphy analytic algorithm
* Current symptoms or history during the past year of Rapid Eye Movement Behavior Disorder or sleep-related violent behavior
* Probable Major Depression, as evidenced by score >10 on the Cornell Scale for Depression in Dementia at Screening
* Unable to tolerate wearing the actigraph. At a minimum, participants must be able to wear the actigraph for 5 complete days out of 7 days' data. A day will be considered complete as long as data from 90% of the 24-hour period are able to be scored.
* Excessive caffeine use that in the opinion of the investigator contributes to the participant's Irregular Sleep-Wake Rhythm Disorder (ISWRD)
* History of drug or alcohol dependency or abuse within approximately the previous 2 years
* Reports habitually consuming more than 14 drinks containing alcohol per week or habitually consumes alcohol within 3 hours before bedtime and unwilling to limit alcohol intake to 2 or fewer drinks per day or forego having alcohol within 3 hours before bedtime for the duration of his/her participation in the study
* Known to be human immunodeficiency virus positive
* Active viral hepatitis (B or C) as demonstrated by positive serology at Screening
* A prolonged QTcF interval (QTcF >450 milliseconds[ms]) as demonstrated by a repeated electrocardiogram (ECG) at Screening (repeated only if initial ECG indicates a QTcF interval >450 ms) (participants with evidence of bundle branch block are not excluded if the block is not clinically significant, as documented by the investigator in the source document)
* Current evidence of clinically significant disease that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments
* Any history of a medical or psychiatric condition other than Alzheimer's Disease dementia that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments
* History of malignancy within the previous 5 years except for adequately treated basal cell or squamous cell skin cancer or cervical carcinoma in situ
* Any suicidal ideation with intent with or without a plan, at the time of or within 6 months of Screening, as indicated by answering "Yes" to questions 4 and 5 on the Suicidal Ideation section of the electronic version of the Columbia Suicide Severity Rating Scale (eC-SSRS)
* Any suicidal behavior within the past 10 years based on the eC-SSRS
* History of violence toward the caregiver or others
* Scheduled for surgery using general anesthesia during the study
* Used any prohibited prescription or over-the-counter concomitant medications within 1 week or 5 half-lives, whichever is longer, before starting actigraphy during Screening
* Used any modality of treatment for ISWRD between Screening and Randomization based on approaches related to circadian rhythms, including phototherapy (light therapy), melatonin and melatonin agonists
* Failed treatment with Belsomra (efficacy and/or safety) following treatment with an appropriate dose and of adequate duration in the opinion of the investigator
* Transmeridian travel across more than 3 time zones between Screening and Randomization, or plans to travel across more than 3 time zones during the study
* Hypersensitivity to lemborexant or to its excipients
* Currently enrolled in another clinical trial, except for observational studies with no treatment component
* Used any investigational drug or device before informed consent (ie, within 30 days or 5× the investigational drug half-life whichever is longer or 6 months for potential disease-modifying drugs)
* Previously participated in any clinical trial of lemborexant

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2020-04-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (46):
- United States (35):
  - Facility #1, Little Rock, Arkansas
  - Facility #1, Rogers, Arkansas
  - Facility #1, Costa Mesa, California
  - Facility #1, Fullerton, California
  - Facility #1, Glendale, California
  - Facility #1, Irvine, California
  - Facility #1, La Jolla, California
  - Facility #1, San Diego, California
  - Facility #1, Santa Monica, California
  - Facility #1, Bradenton, Florida
  - Facility #1, Brandon, Florida
  - Facility #1, Brooksville, Florida
  - Facility #1, Hallandale, Florida
  - Facility #1, Miami, Florida
  - Facility #1, Miami Lakes, Florida
  - Facility #1, Miami Springs, Florida
  - Facility #1, Orlando, Florida
  - Facility #2, Orlando, Florida
  - Facility #1, Sunrise, Florida
  - Facility #2, Tampa, Florida
  - Facility #1, Atlanta, Georgia
  - Facility #1, Columbus, Georgia
  - Facility #1, Macon, Georgia
  - Facility #1, Wichita, Kansas
  - Facility #1, Belmont, Massachusetts
  - Nevada Senior Services (NSS) Adult Day Care Center, Henderson, Nevada
  - Facility #1, Las Vegas, Nevada
  - Facility #1, Toms River, New Jersey
  - Facility #2, Toms River, New Jersey
  - Facility #1, Charlotte, North Carolina
  - Facility #2, Durham, North Carolina
  - Facility #1, Raleigh, North Carolina
  - Facility #1, Norristown, Pennsylvania
  - Facility #1, Willow Grove, Pennsylvania
  - Facility #1, Columbia, South Carolina
- Japan (8):
  - Eisai Trial Site #1, Nagoya, Aichi-ken
  - Eisai Trial Site #1, Fujisawa, Kanagawa
  - Eisai Trial Site #1, Kawasaki-shi, Kanagawa
  - Eisai Trial Site #1, Wako, Saitama
  - Eisai Trial Site #1, Kodaira, Tokyo
  - Eisai Trial Site #1, Setagaya City, Tokyo
  - Eisai Trial Site #1, Shinjuku, Tokyo
  - Eisai Trial Site #1, Tachikawa-shi, Tokyo
- United Kingdom (3):
  - Brighton and Sussex Medical School, Brighton, East Sussex
  - Cognitive Treatment and Research Unit, Crowborough, East Sussex
  - University of Edinburgh - PPDS, Edinburgh

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 57 investigative sites in the United States, Japan and United Kingdom from 20 Dec 2016 to 17 Apr 2020.
Pre-assignment Details: In Core phase, a total of 214 participants were screened, of which 151 were screen failures and 63 were randomized and enrolled in to the study. Of these 63 participants, 62 received the study treatment (1 participant was inadvertently randomized but did not receive any study drug). In Extension phase, a total of 25 participants who completed the Core Phase, gave consent to join Extension phase were enrolled and treated.
Groups:
- Core Phase: Lemborexant-matched Placebo: Participants received two lemborexant-matched placebo, tablets, orally, once daily, immediately (within 5 minutes) before the bedtime at night for 28 consecutive nights in 4-week treatment period.
- Core Phase: Lemborexant 2.5 mg: Participants received one lemborexant 2.5 milligrams (mg) and one lemborexant-matched placebo, tablets, orally, once daily, immediately (within 5 minutes) before the bedtime at night for 28 consecutive nights in 4-week treatment period.
- Core Phase: Lemborexant 5 mg: Participants received one lemborexant 5 mg and one lemborexant-matched placebo, tablets, orally, once daily, immediately (within 5 minutes) before the bedtime at night for 28 consecutive nights in 4-week treatment period.
- Core Phase: Lemborexant 10 mg: Participants received one lemborexant 10 mg and one lemborexant-matched placebo, tablets, orally, once daily, immediately (within 5 minutes) before the bedtime at night for 28 consecutive nights in 4-week treatment period.
- Core Phase: Lemborexant 15 mg: Participants received one lemborexant 5 mg and one lemborexant 10 mg, tablets, orally, once daily, immediately (within 5 minutes) before the bedtime at night for 28 consecutive nights in 4-week treatment period.
- Extension Phase: Lemborexant 5 mg: Participants who completed the core study end of study (EOS) visit within 30 days prior to enrollment in extension phase were eligible to participate in extension phase. Participants received one lemborexant 5 mg, tablet, orally, once daily, immediately (within 5 minutes) before the bedtime at night until lemborexant is commercially available, or until the lemborexant clinical development program for Irregular Sleep-Wake Rhythm Disorder (ISWRD) is discontinued or up to 30 months.
- Extension Phase: Lemborexant 10 mg: Participants who completed the core study EOS visit within 30 days prior to enrollment in extension phase were eligible to participate in extension phase. Participants received one lemborexant 10 mg, tablet, orally, once daily, immediately (within 5 minutes) before the bedtime at night until lemborexant is commercially available, or until the lemborexant clinical development program for ISWRD is discontinued or up to 30 months.
- Extension Phase: Lemborexant 15 mg: Participants who completed the core study EOS visit within 30 days prior to enrollment in extension phase were eligible to participate in extension phase. Participants received one lemborexant 5 mg and one lemborexant 10 mg, tablets, orally, once daily, immediately (within 5 minutes) before the bedtime at night until lemborexant is commercially available, or until the lemborexant clinical development program for ISWRD is discontinued or up to 30 months.
Period: Core Phase
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg | Extension Phase: Lemborexant 5 mg | Extension Phase: Lemborexant 10 mg | Extension Phase: Lemborexant 15 mg
Started | 12 | 12 | 14 | 13 | 12 | 0 | 0 | 0
Treated | 12 | 12 | 13 | 13 | 12 | 0 | 0 | 0
Completed | 12 | 12 | 13 | 13 | 12 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized but not treated | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Extension Phase
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg | Extension Phase: Lemborexant 5 mg | Extension Phase: Lemborexant 10 mg | Extension Phase: Lemborexant 15 mg
Started | 0 | 0 | 0 | 0 | 0 | 5 | 14 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 5 | 14 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Administrative Reason | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3
Not completed — Loss of caregiver | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Others | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included the group of randomized participants who received at least 1 dose of randomized study drug and had at least 1 postdose safety assessment.
Groups:
- Core Phase: Lemborexant 2.5 mg: Participants received one lemborexant 2.5 mg and one lemborexant-matched placebo, tablets, orally, once daily, immediately (within 5 minutes) before the bedtime at night for 28 consecutive nights in 4-week treatment period.
- Total: Total of all reporting groups
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg | Total
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.3 (6.15) | 76.5 (6.32) | 76.9 (7.98) | 71.8 (7.05) | 71.9 (6.11) | 74.5 (6.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 8 | 6 | 10 | 37
  Male | 5 | 6 | 5 | 7 | 2 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 4 | 6 | 8 | 24
  Not Hispanic or Latino | 8 | 10 | 9 | 7 | 4 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 2 | 3 | 2 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 1 | 1 | 7
  White | 8 | 9 | 8 | 9 | 9 | 43
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Core Phase: Change From Baseline in Mean Actigraphy Sleep Efficiency (aSE) With Lemborexant Compared to Placebo During Week 1 of Treatment
Description: aSE was defined as the percentage of time spent in bed nocturnal sleeping, as measured by actigraphy. Sleep efficiency was calculated as the total duration of sleep epochs during the predefined 8-hour nocturnal sleep period divided by 8 hours and multiplied by 100. Higher values were better. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average first 7 nights of treatment was reported.
Time Frame: Baseline, Week 1
Population: The full analysis set (FAS) included group of randomized participants who received at least 1 dose of randomized study drug and had at least 1 postdose efficacy measurement. Participants who were evaluable for this measure at given time point were included for the assessment.
Measure: Mean (Standard Deviation); unit: percentage of sleep time
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
percentage of sleep time
  Baseline | 76.34 (6.559) | 77.64 (7.883) | 78.45 (6.844) | 76.38 (8.037) | 77.35 (8.624)
  Change at Week 1: number analyzed (Participants) | 12 | 11 | 13 | 13 | 12
  Change at Week 1 | 0.14 (5.766) | 2.43 (3.910) | 3.87 (4.646) | -0.17 (5.861) | 0.05 (4.475)

2. Primary Outcome: Core Phase: Change From Baseline in Mean aSE With Lemborexant Compared to Placebo During Week 2 of Treatment
Description: aSE was defined as the percentage of time spent in bed nocturnal sleeping, as measured by actigraphy. Sleep efficiency was calculated as the total duration of sleep epochs during the predefined 8-hour nocturnal sleep period divided by 8 hours and multiplied by 100. Higher values were better. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average second 7 nights of treatment was reported.
Time Frame: Baseline, Week 2
Population: The FAS included group of randomized participants who received at least 1 dose of randomized study drug and had at least 1 postdose efficacy measurement. Participants who were evaluable for this measure at given time point were included for the assessment.
Measure: Mean (Standard Deviation); unit: percentage of sleep time
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
percentage of sleep time
  Baseline | 76.34 (6.559) | 77.64 (7.883) | 78.45 (6.844) | 76.38 (8.037) | 77.35 (8.624)
  Change at Week 2: number analyzed (Participants) | 12 | 10 | 13 | 13 | 12
  Change at Week 2 | -1.31 (7.004) | 2.17 (2.833) | 1.65 (4.644) | -1.41 (5.896) | -0.07 (5.449)

3. Primary Outcome: Core Phase: Change From Baseline in Mean aSE With Lemborexant Compared to Placebo During Week 3 of Treatment
Description: aSE was defined as the percentage of time spent in bed nocturnal sleeping, as measured by actigraphy. Sleep efficiency was calculated as the total duration of sleep epochs during the predefined 8-hour nocturnal sleep period divided by 8 hours and multiplied by 100. Higher values were better. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average third 7 nights of treatment was reported.
Time Frame: Baseline, Week 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of sleep time
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
percentage of sleep time
  Baseline | 76.34 (6.559) | 77.64 (7.883) | 78.45 (6.844) | 76.38 (8.037) | 77.35 (8.624)
  Change at Week 3: number analyzed (Participants) | 11 | 11 | 12 | 12 | 12
  Change at Week 3 | -0.30 (10.552) | 1.68 (3.229) | 0.91 (7.571) | -1.49 (4.442) | 1.10 (7.112)

4. Primary Outcome: Core Phase: Change From Baseline in Mean aSE With Lemborexant Compared to Placebo During Week 4 of Treatment
Description: aSE was defined as the percentage of time spent in bed nocturnal sleeping, as measured by actigraphy. Sleep efficiency was calculated as the total duration of sleep epochs during the predefined 8-hour nocturnal sleep period divided by 8 hours and multiplied by 100. Higher values were better. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average last 7 nights of treatment was reported.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of sleep time
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
percentage of sleep time
  Baseline | 76.34 (6.559) | 77.64 (7.883) | 78.45 (6.844) | 76.38 (8.037) | 77.35 (8.624)
  Change at Week 4: number analyzed (Participants) | 11 | 11 | 12 | 11 | 12
  Change at Week 4 | -0.78 (9.555) | 1.68 (4.696) | 0.00 (5.547) | -1.04 (5.920) | -0.81 (7.735)
Statistical Analysis 1: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 2.5 mg; Test type: Superiority; p = 0.1099, MMRM — Based on a mixed model for repeated measure (MMRM) analysis adjusted for baseline value, country, visit and treatment by visit interaction; Least square mean (LSM) difference = 3.177, 95% CI 2-sided [-0.741 to 7.096]
Statistical Analysis 2: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 5 mg; Test type: Superiority; p = 0.1576, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 2.802, 95% CI 2-sided [-1.119 to 6.723]
Statistical Analysis 3: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.6160, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -0.960, 95% CI 2-sided [-4.777 to 2.857]
Statistical Analysis 4: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 15 mg; Test type: Superiority; p = 0.7135, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 0.713, 95% CI 2-sided [-3.160 to 4.585]

5. Primary Outcome: Core Phase: Change From Baseline in Mean Sleep Fragmentation Index (SFI) During Week 1 of Treatment
Description: The SFI was defined as the sum of a movement index (MI) and a fragmentation index (FI) during the logged sleep period. The MI was equal to the epochs of wake per time in bed (TBI) multiplied by 100. The FI was equal to the number of less than or equal to (<=) 1-minute periods of immobility/total number of periods of immobility of all durations during the defined nocturnal sleep period multiplied by 100. Value ranges from 0-100 percent (%) (lower values were better). SFI was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average first 7 nights of treatment was reported.
Time Frame: Baseline, Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of immobile bouts
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
percentage of immobile bouts
  Baseline | 58.51 (12.923) | 53.87 (17.594) | 50.07 (12.493) | 54.75 (16.380) | 54.78 (15.338)
  Change at Week 1: number analyzed (Participants) | 12 | 11 | 13 | 12 | 12
  Change at Week 1 | -1.43 (9.294) | -5.80 (11.388) | -8.16 (8.802) | -2.55 (11.756) | -3.52 (8.882)

6. Primary Outcome: Core Phase: Change From Baseline in Mean SFI During Week 2 of Treatment
Description: The SFI was defined as the sum of a MI and a FI during the logged sleep period. The MI was equal to the epochs of wake per TBI multiplied by 100. The FI was equal to the number <=1-minute periods of immobility/total number of periods of immobility of all durations during the defined nocturnal sleep period multiplied by 100. Value ranges from 0-100% (lower values were better). SFI was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average second 7 nights of treatment was reported.
Time Frame: Baseline, Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of immobile bouts
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
percentage of immobile bouts
  Baseline | 58.51 (12.923) | 53.87 (17.594) | 50.07 (12.493) | 54.75 (16.380) | 54.78 (15.338)
  Change at Week 2: number analyzed (Participants) | 12 | 10 | 13 | 13 | 12
  Change at Week 2 | 2.52 (11.845) | -6.91 (5.994) | -4.95 (8.399) | 0.34 (14.194) | -3.18 (8.971)

7. Primary Outcome: Core Phase: Change From Baseline in Mean SFI During Week 3 of Treatment
Description: The SFI was defined as the sum of a MI and a FI during the logged sleep period. The MI was equal to the epochs of wake per TBI multiplied by 100. The FI was equal to the number <=1-minute periods of immobility/total number of periods of immobility of all durations during the defined nocturnal sleep period multiplied by 100. Value ranges from 0-100% (lower values were better). SFI was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average third 7 nights of treatment was reported.
Time Frame: Baseline, Week 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of immobile bouts
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
percentage of immobile bouts
  Baseline | 58.51 (12.923) | 53.87 (17.594) | 50.07 (12.493) | 54.75 (16.380) | 54.78 (15.338)
  Change at Week 3: number analyzed (Participants) | 11 | 11 | 12 | 12 | 12
  Change at Week 3 | -3.30 (18.512) | -2.79 (7.541) | -5.22 (11.974) | 0.36 (9.018) | -4.92 (9.572)

8. Primary Outcome: Core Phase: Change From Baseline in Mean SFI During Week 4 of Treatment
Description: The SFI was defined as the sum of a MI and a FI during the logged sleep period. The MI was equal to the epochs of wake per TBI multiplied by 100. The FI was equal to the number <=1-minute periods of immobility/total number of periods of immobility of all durations during the defined nocturnal sleep period multiplied by 100. Value ranges from 0-100% (lower values were better). SFI was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average last 7 nights of treatment was reported.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of immobile bouts
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
percentage of immobile bouts
  Baseline | 58.51 (12.923) | 53.87 (17.594) | 50.07 (12.493) | 54.75 (16.380) | 54.78 (15.338)
  Change at Week 4: number analyzed (Participants) | 11 | 11 | 12 | 11 | 12
  Change at Week 4 | -1.39 (19.383) | -1.35 (8.821) | -1.96 (8.459) | -0.45 (13.389) | -1.68 (12.683)
Statistical Analysis 1: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 2.5 mg; Test type: Superiority; p = 0.1582, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -5.098, 95% CI 2-sided [-12.240 to 2.045]
Statistical Analysis 2: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 5 mg; Test type: Superiority; p = 0.0961, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -6.105, 95% CI 2-sided [-13.332 to 1.122]
Statistical Analysis 3: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.8449, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 0.680, 95% CI 2-sided [-6.262 to 7.623]
Statistical Analysis 4: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 15 mg; Test type: Superiority; p = 0.3747, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -3.140, 95% CI 2-sided [-10.178 to 3.897]

9. Primary Outcome: Core Phase: Change From Baseline in the Mean Duration of Wake Bouts (aMeanDurWB) During Week 1 of Treatment
Description: aMeanDurWB was defined as an average duration of all wake bouts that occurred during the defined nocturnal predefined sleep period. The wake bout was defined as continuous wake of 10 minutes or longer. Lower values were better. aMeanDurWB was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average first 7 nights of treatment was reported.
Time Frame: Baseline, Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
minutes
  Baseline | 20.32 (6.625) | 20.40 (5.140) | 20.62 (5.898) | 21.89 (4.885) | 21.94 (7.790)
  Change at Week 1: number analyzed (Participants) | 12 | 11 | 13 | 12 | 12
  Change at Week 1 | -1.65 (5.078) | -1.99 (2.825) | -0.51 (6.522) | -0.82 (5.722) | 1.54 (5.378)

10. Primary Outcome: Core Phase: Change From Baseline in the aMeanDurWB During Week 2 of Treatment
Description: aMeanDurWB was defined as an average duration of all wake bouts that occurred during the defined nocturnal predefined sleep period. The wake bout was defined as continuous wake of 10 minutes or longer. Lower values were better. aMeanDurWB was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average second 7 nights of treatment was reported.
Time Frame: Baseline, Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
minutes
  Baseline | 20.32 (6.625) | 20.40 (5.140) | 20.62 (5.898) | 21.89 (4.885) | 21.94 (7.790)
  Change at Week 2: number analyzed (Participants) | 12 | 10 | 13 | 12 | 12
  Change at Week 2 | -0.32 (7.904) | 1.79 (12.957) | 4.71 (13.845) | 1.54 (6.333) | 2.57 (6.708)

11. Primary Outcome: Core Phase: Change From Baseline in the aMeanDurWB During Week 3 of Treatment
Description: aMeanDurWB was defined as an average duration of all wake bouts that occurred during the defined nocturnal predefined sleep period. The wake bout was defined as continuous wake of 10 minutes or longer. Lower values were better. aMeanDurWB was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average third 7 nights of treatment was reported.
Time Frame: Baseline, Week 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
minutes
  Baseline | 20.32 (6.625) | 20.40 (5.140) | 20.62 (5.898) | 21.89 (4.885) | 21.94 (7.790)
  Change at Week 3: number analyzed (Participants) | 11 | 11 | 11 | 12 | 12
  Change at Week 3 | -2.88 (7.928) | 3.67 (7.833) | -0.52 (4.595) | -0.64 (5.482) | 2.76 (7.489)

12. Primary Outcome: Core Phase: Change From Baseline in the aMeanDurWB During Week 4 of Treatment
Description: aMeanDurWB was defined as an average duration of all wake bouts that occurred during the defined nocturnal predefined sleep period. The wake bout was defined as continuous wake of 10 minutes or longer. Lower values were better. aMeanDurWB was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average last 7 nights of treatment was reported.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
minutes
  Baseline | 20.32 (6.625) | 20.40 (5.140) | 20.62 (5.898) | 21.89 (4.885) | 21.94 (7.790)
  Change at Week 4: number analyzed (Participants) | 11 | 11 | 11 | 11 | 12
  Change at Week 4 | -1.26 (8.621) | -0.43 (8.053) | 3.16 (8.140) | -2.03 (4.947) | 3.38 (12.354)
Statistical Analysis 1: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 2.5 mg; Test type: Superiority; p = 0.3966, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 1.932, 95% CI 2-sided [-2.601 to 6.465]
Statistical Analysis 2: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 5 mg; Test type: Superiority; p = 0.1381, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 3.386, 95% CI 2-sided [-1.125 to 7.897]
Statistical Analysis 3: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.5487, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 1.337, 95% CI 2-sided [-3.104 to 5.778]
Statistical Analysis 4: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 15 mg; Test type: Superiority; p = 0.0581, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 4.320, 95% CI 2-sided [-0.153 to 8.793]

13. Primary Outcome: Core Phase: Change From Baseline in Mean Actigraphy Wake Efficiency (aWE) During Week 1 of Treatment
Description: aWE was defined as the percentage of time spent awake in bed during defined wake period, as measured by actigraphy. Wake efficiency was calculated as the total duration of wake epochs during 16 hours outside of the predefined sleep period divided by 16 hours and multiplied by 100. Higher values were better. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average first 7 nights of treatment was reported.
Time Frame: Baseline, Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of wake time
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
percentage of wake time
  Baseline | 69.74 (12.609) | 70.57 (11.669) | 72.53 (11.473) | 67.19 (11.523) | 70.67 (11.221)
  Change at Week 1: number analyzed (Participants) | 12 | 11 | 13 | 12 | 12
  Change at Week 1 | 0.59 (4.177) | -2.41 (6.726) | 1.09 (6.793) | -1.55 (9.216) | -2.37 (8.779)

14. Primary Outcome: Core Phase: Change From Baseline in Mean aWE During Week 2 of Treatment
Description: aWE was defined as the percentage of time spent awake in bed during defined wake period, as measured by actigraphy. Wake efficiency was calculated as the total duration of wake epochs during 16 hours outside of the predefined sleep period divided by 16 hours and multiplied by 100. Higher values were better. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average second 7 nights of treatment was reported.
Time Frame: Baseline, Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of wake time
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
percentage of wake time
  Baseline | 69.74 (12.609) | 70.57 (11.669) | 72.53 (11.473) | 67.19 (11.523) | 70.67 (11.221)
  Change at Week 2: number analyzed (Participants) | 12 | 10 | 13 | 12 | 12
  Change at Week 2 | 2.14 (2.773) | -1.54 (6.550) | 1.04 (7.511) | -3.16 (12.816) | -0.63 (5.617)

15. Primary Outcome: Core Phase: Change From Baseline in Mean aWE During Week 3 of Treatment
Description: aWE was defined as the percentage of time spent awake in bed during defined wake period, as measured by actigraphy. Wake efficiency was calculated as the total duration of wake epochs during 16 hours outside of the predefined sleep period divided by 16 hours and multiplied by 100. Higher values were better. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average third 7 nights of treatment was reported.
Time Frame: Baseline, Week 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of wake time
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
percentage of wake time
  Baseline | 69.74 (12.609) | 70.57 (11.669) | 72.53 (11.473) | 67.19 (11.523) | 70.67 (11.221)
  Change at Week 3: number analyzed (Participants) | 11 | 11 | 12 | 12 | 12
  Change at Week 3 | 1.64 (5.451) | -2.37 (6.239) | 2.34 (8.370) | -4.99 (11.479) | -1.83 (5.579)

16. Primary Outcome: Core Phase: Change From Baseline in Mean aWE During Week 4 of Treatment
Description: aWE was defined as the percentage of time spent awake in bed during defined wake period, as measured by actigraphy. Wake efficiency was calculated as the total duration of wake epochs during 16 hours outside of the predefined sleep period divided by 16 hours and multiplied by 100. Higher values were better. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average last 7 nights of treatment was reported.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of wake time
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
percentage of wake time
  Baseline | 69.74 (12.609) | 70.57 (11.669) | 72.53 (11.473) | 67.19 (11.523) | 70.67 (11.221)
  Change at Week 4: number analyzed (Participants) | 11 | 11 | 12 | 11 | 12
  Change at Week 4 | 2.03 (6.841) | -2.29 (7.724) | 3.62 (8.586) | -2.65 (9.627) | -0.43 (5.848)
Statistical Analysis 1: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 2.5 mg; Test type: Superiority; p = 0.1777, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -3.437, 95% CI 2-sided [-8.481 to 1.608]
Statistical Analysis 2: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 5 mg; Test type: Superiority; p = 0.5630, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 1.458, 95% CI 2-sided [-3.564 to 6.479]
Statistical Analysis 3: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.0482, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -4.994, 95% CI 2-sided [-9.946 to -0.041]
Statistical Analysis 4: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 15 mg; Test type: Superiority; p = 0.3036, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -2.593, 95% CI 2-sided [-7.599 to 2.413]

17. Primary Outcome: Core Phase: Change From Baseline in Mean Wake Fragmentation Index (WFI) During Week 1 of Treatment
Description: The WFI were calculated as the sum of an immobility index (II) and a FI during the logged wake period. The II was equal to the epochs of immobility per the 16 hours outside of the defined sleep period multiplied by 100. The FI was equal to the number of <=1-minute periods of mobility/total number of periods of mobility the 16 hours outside of the defined sleep period multiplied by 100. Value ranges from 0-100 percent (lower values were better). The WFI was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average first 7 nights of treatment was reported.
Time Frame: Baseline, Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of immobile bouts
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
percentage of immobile bouts
  Baseline | 92.43 (18.547) | 85.72 (16.137) | 86.53 (18.705) | 94.76 (17.262) | 87.96 (15.928)
  Change at Week 1: number analyzed (Participants) | 12 | 11 | 13 | 12 | 12
  Change at Week 1 | -0.14 (6.968) | 4.22 (9.988) | -2.18 (10.571) | 2.01 (13.017) | 3.25 (13.006)

18. Primary Outcome: Core Phase: Change From Baseline in Mean WFI During Week 2 of Treatment
Description: The WFI were calculated as the sum of an II and a FI during the logged wake period. The II was equal to the epochs of immobility per the 16 hours outside of the defined sleep period multiplied by 100. The FI was equal to the number of <=1-minute periods of mobility/total number of periods of mobility the 16 hours outside of the defined sleep period multiplied by 100. Value ranges from 0-100% (lower values were better). The WFI was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average second 7 nights of treatment was reported.
Time Frame: Baseline, Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of immobile bouts
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
percentage of immobile bouts
  Baseline | 92.43 (18.547) | 85.72 (16.137) | 86.53 (18.705) | 94.76 (17.262) | 87.96 (15.928)
  Change at Week 2 | -3.76 (3.940) | 4.12 (8.671) | -2.36 (11.453) | 5.09 (19.006) | 1.78 (9.271)

19. Primary Outcome: Core Phase: Change From Baseline in Mean WFI During Week 3 of Treatment
Description: The WFI were calculated as the sum of an II and a FI during the logged wake period. The II was equal to the epochs of immobility per the 16 hours outside of the defined sleep period multiplied by 100. The FI was equal to the number of <=1-minute periods of mobility/total number of periods of mobility the 16 hours outside of the defined sleep period multiplied by 100. Value ranges from 0-100% (lower values were better). The WFI was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average third 7 nights of treatment was reported.
Time Frame: Baseline, Week 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of immobile bouts
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
percentage of immobile bouts
  Baseline | 92.43 (18.547) | 85.72 (16.137) | 86.53 (18.705) | 94.76 (17.262) | 87.96 (15.928)
  Change at Week 3: number analyzed (Participants) | 11 | 11 | 12 | 12 | 12
  Change at Week 3 | -1.65 (7.980) | 4.70 (9.674) | -3.69 (13.236) | 6.88 (16.704) | 2.10 (8.631)

20. Primary Outcome: Core Phase: Change From Baseline in Mean WFI During Week 4 of Treatment
Description: The WFI were calculated as the sum of an II and a FI during the logged wake period. The II was equal to the epochs of immobility per the 16 hours outside of the defined sleep period multiplied by 100. The FI was equal to the number of <=1-minute periods of mobility/total number of periods of mobility the 16 hours outside of the defined sleep period multiplied by 100. Value ranges from 0-100% (lower values were better). The WFI was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average last 7 nights of treatment was reported.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of immobile bouts
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
percentage of immobile bouts
  Baseline | 92.43 (18.547) | 85.72 (16.137) | 86.53 (18.705) | 94.76 (17.262) | 87.96 (15.928)
  Change at Week 4: number analyzed (Participants) | 11 | 11 | 12 | 11 | 12
  Change at Week 4 | -3.01 (10.620) | 4.55 (10.930) | -6.93 (14.428) | 2.77 (13.407) | 1.22 (8.054)
Statistical Analysis 1: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 2.5 mg; Test type: Superiority; p = 0.1991, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 4.845, 95% CI 2-sided [-2.624 to 12.313]
Statistical Analysis 2: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 5 mg; Test type: Superiority; p = 0.2982, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -3.872, 95% CI 2-sided [-11.263 to 3.518]
Statistical Analysis 3: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.0664, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 6.776, 95% CI 2-sided [-0.474 to 14.025]
Statistical Analysis 4: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 15 mg; Test type: Superiority; p = 0.4148, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 3.017, 95% CI 2-sided [-4.344 to 10.379]

21. Primary Outcome: Core Phase: Change From Baseline in the Mean Duration of Sleep Bouts (aMeanDurSB) During Week 1 of Treatment
Description: aMeanDurSB was defined as an average duration of all sleep bouts that occurred during the 16 hours outside of the predefined nocturnal sleep period. The sleep bout was defined as the continuous sleep of 10 minutes or longer. Lower values were better. aMeanDurSB was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average first 7 nights of treatment was reported.
Time Frame: Baseline, Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
minutes
  Baseline | 18.36 (4.620) | 20.65 (3.638) | 23.13 (5.919) | 19.84 (3.364) | 23.30 (10.862)
  Change at Week 1: number analyzed (Participants) | 12 | 11 | 13 | 12 | 12
  Change at Week 1 | 2.15 (2.539) | 0.09 (4.056) | -1.12 (5.202) | -0.40 (3.394) | -3.19 (10.405)

22. Primary Outcome: Core Phase: Change From Baseline in the aMeanDurSB During Week 2 of Treatment
Description: aMeanDurSB was defined as an average duration of all sleep bouts that occurred during the 16 hours outside of the predefined nocturnal sleep period. The sleep bout was defined as the continuous sleep of 10 minutes or longer. Lower values were better. aMeanDurSB was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average second 7 nights of treatment was reported.
Time Frame: Baseline, Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
minutes
  Baseline | 18.36 (4.620) | 20.65 (3.638) | 23.13 (5.919) | 19.84 (3.364) | 23.30 (10.862)
  Change at Week 2: number analyzed (Participants) | 12 | 10 | 13 | 12 | 12
  Change at Week 2 | 0.25 (2.999) | -0.88 (4.679) | -2.52 (5.965) | -0.80 (2.961) | -3.95 (8.980)

23. Primary Outcome: Core Phase: Change From Baseline in the aMeanDurSB During Week 3 of Treatment
Description: aMeanDurSB was defined as an average duration of all sleep bouts that occurred during the 16 hours outside of the predefined nocturnal sleep period. The sleep bout was defined as the continuous sleep of 10 minutes or longer. Lower values were better. aMeanDurSB was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average third 7 nights of treatment was reported.
Time Frame: Baseline, Week 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
minutes
  Baseline | 18.36 (4.620) | 20.65 (3.638) | 23.13 (5.919) | 19.84 (3.364) | 23.30 (10.862)
  Change at Week 3: number analyzed (Participants) | 11 | 11 | 12 | 12 | 12
  Change at Week 3 | -0.14 (3.249) | -1.17 (4.056) | -3.80 (3.701) | -0.68 (2.292) | -4.15 (10.264)

24. Primary Outcome: Core Phase: Change From Baseline in the aMeanDurSB During Week 4 of Treatment
Description: aMeanDurSB was defined as an average duration of all sleep bouts that occurred during the 16 hours outside of the predefined nocturnal sleep period. The sleep bout was defined as the continuous sleep of 10 minutes or longer. Lower values were better. aMeanDurSB was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average last 7 nights of treatment was reported.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
minutes
  Baseline | 18.36 (4.620) | 20.65 (3.638) | 23.13 (5.919) | 19.84 (3.364) | 23.30 (10.862)
  Change at Week 4: number analyzed (Participants) | 11 | 11 | 12 | 11 | 12
  Change at Week 4 | 1.00 (4.568) | -1.31 (3.639) | -2.80 (5.727) | -0.03 (2.307) | -5.30 (9.745)
Statistical Analysis 1: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 2.5 mg; Test type: Superiority; p = 0.9599, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 0.063, 95% CI 2-sided [-2.452 to 2.579]
Statistical Analysis 2: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 5 mg; Test type: Superiority; p = 0.8541, MMRM — Based on a MMRM analysis adjusted for baseline value, country, Visit and treatment by Visit interaction; LSM Difference = -0.238, 95% CI 2-sided [-2.817 to 2.342]
Statistical Analysis 3: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.8117, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -0.293, 95% CI 2-sided [-2.745 to 2.160]
Statistical Analysis 4: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 15 mg; Test type: Superiority; p = 0.2274, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -1.557, 95% CI 2-sided [-4.113 to 1.000]

25. Primary Outcome: Core Phase: Change From Baseline in Mean Intradaily Variability Over Week 1 of Treatment
Description: Intradaily variability gives an indication of irregular sleep-wake rhythm disorder (ISWRD) by quantifying the number and strength of transitions between rest and activity bouts, derived by the ratio of the mean squares of the difference between all successive hours (first derivative) and the mean squares around the grand mean (overall variance). The variable has a theoretical range of 0 to 2, with higher values indicating higher fragmentation. Intradaily variability was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average first 7 nights of treatment was reported.
Time Frame: Baseline, Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
ratio
  Baseline | 1.10 (0.262) | 0.90 (0.272) | 0.98 (0.295) | 1.10 (0.295) | 1.03 (0.330)
  Change at Week 1: number analyzed (Participants) | 12 | 11 | 13 | 11 | 12
  Change at Week 1 | -0.01 (0.200) | 0.06 (0.218) | -0.03 (0.237) | 0.10 (0.271) | -0.01 (0.278)

26. Primary Outcome: Core Phase: Change From Baseline in Mean Intradaily Variability Over Week 2 of Treatment
Description: Intradaily variability gives an indication of ISWRD by quantifying the number and strength of transitions between rest and activity bouts, derived by the ratio of the mean squares of the difference between all successive hours (first derivative) and the mean squares around the grand mean (overall variance). The variable has a theoretical range of 0 to 2, with higher values indicating higher fragmentation. Intradaily variability was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average second 7 nights of treatment was reported.
Time Frame: Baseline, Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
ratio
  Baseline | 1.10 (0.262) | 0.90 (0.272) | 0.98 (0.295) | 1.10 (0.295) | 1.03 (0.330)
  Change at Week 2: number analyzed (Participants) | 12 | 9 | 12 | 12 | 11
  Change at Week 2 | -0.05 (0.132) | 0.14 (0.325) | 0.02 (0.235) | 0.07 (0.143) | 0.05 (0.234)

27. Primary Outcome: Core Phase: Change From Baseline in Mean Intradaily Variability Over Week 3 of Treatment
Description: Intradaily variability gives an indication of ISWRD by quantifying the number and strength of transitions between rest and activity bouts, derived by the ratio of the mean squares of the difference between all successive hours (first derivative) and the mean squares around the grand mean (overall variance). The variable has a theoretical range of 0 to 2, with higher values indicating higher fragmentation. Intradaily variability was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average third 7 nights of treatment was reported.
Time Frame: Baseline, Week 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
ratio
  Baseline | 1.10 (0.262) | 0.90 (0.272) | 0.98 (0.295) | 1.10 (0.295) | 1.03 (0.330)
  Change at Week 3: number analyzed (Participants) | 11 | 11 | 12 | 12 | 12
  Change at Week 3 | -0.06 (0.243) | 0.07 (0.246) | -0.00 (0.241) | -0.06 (0.311) | -0.01 (0.219)

28. Primary Outcome: Core Phase: Change From Baseline in Mean Intradaily Variability Over Week 4 of Treatment
Description: Intradaily variability gives an indication of ISWRD by quantifying the number and strength of transitions between rest and activity bouts, derived by the ratio of the mean squares of the difference between all successive hours (first derivative) and the mean squares around the grand mean (overall variance). The variable has a theoretical range of 0 to 2, with higher values indicating higher fragmentation. Intradaily variability was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average last 7 nights of treatment was reported.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
ratio
  Baseline | 1.10 (0.262) | 0.90 (0.272) | 0.98 (0.295) | 1.10 (0.295) | 1.03 (0.330)
  Change at Week 4: number analyzed (Participants) | 7 | 10 | 8 | 8 | 9
  Change at Week 4 | -0.10 (0.324) | 0.10 (0.196) | 0.02 (0.157) | -0.12 (0.274) | -0.10 (0.222)
Statistical Analysis 1: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 2.5 mg; Test type: Superiority; p = 0.2421, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 0.086, 95% CI 2-sided [-0.060 to 0.232]
Statistical Analysis 2: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 5 mg; Test type: Superiority; p = 0.8661, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -0.012, 95% CI 2-sided [-0.155 to 0.131]
Statistical Analysis 3: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.4251, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 0.057, 95% CI 2-sided [-0.085 to 0.199]
Statistical Analysis 4: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 15 mg; Test type: Superiority; p = 0.7248, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 0.025, 95% CI 2-sided [-0.116 to 0.166]

29. Primary Outcome: Core Phase: Change From Baseline in Mean Interdaily Stability (IS) Over Week 1 of Treatment
Description: IS gives an indication of the stability of the sleep-wake rhythm across days, and varies from zero (low stability) to 1 (high stability). IS was derived by the ratio between the variance of the average 24-hour pattern around the mean and the overall variance. Higher values indicated stable rhythm. IS was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average first 7 nights of treatment was reported.
Time Frame: Baseline, Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
ratio
  Baseline | 0.45 (0.173) | 0.47 (0.111) | 0.49 (0.118) | 0.46 (0.160) | 0.41 (0.104)
  Change at Week 1: number analyzed (Participants) | 12 | 11 | 13 | 11 | 12
  Change at Week 1 | 0.04 (0.083) | -0.02 (0.089) | 0.04 (0.115) | -0.00 (0.155) | 0.06 (0.063)

30. Primary Outcome: Core Phase: Change From Baseline in Mean IS Over Week 2 of Treatment
Description: IS gives an indication of the stability of the sleep-wake rhythm across days, and varies from zero (low stability) to 1 (high stability). IS was derived by the ratio between the variance of the average 24-hour pattern around the mean and the overall variance. Higher values indicated stable rhythm. IS was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average second 7 nights of treatment was reported.
Time Frame: Baseline, Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
ratio
  Baseline | 0.45 (0.173) | 0.47 (0.111) | 0.49 (0.118) | 0.46 (0.160) | 0.41 (0.104)
  Change at Week 2: number analyzed (Participants) | 12 | 9 | 12 | 12 | 11
  Change at Week 2 | 0.06 (0.093) | -0.01 (0.101) | 0.03 (0.133) | -0.06 (0.091) | 0.09 (0.085)

31. Primary Outcome: Core Phase: Change From Baseline in Mean IS Over Week 3 of Treatment
Description: IS gives an indication of the stability of the sleep-wake rhythm across days, and varies from zero (low stability) to 1 (high stability). IS was derived by the ratio between the variance of the average 24-hour pattern around the mean and the overall variance. Higher values indicated stable rhythm. IS was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average third 7 nights of treatment was reported.
Time Frame: Baseline, Week 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
ratio
  Baseline | 0.45 (0.173) | 0.47 (0.111) | 0.49 (0.118) | 0.46 (0.160) | 0.41 (0.104)
  Change at Week 3: number analyzed (Participants) | 11 | 11 | 12 | 12 | 12
  Change at Week 3 | 0.03 (0.104) | -0.01 (0.107) | 0.03 (0.115) | -0.04 (0.136) | 0.04 (0.075)

32. Primary Outcome: Core Phase: Change From Baseline in Mean IS Over Week 4 of Treatment
Description: IS gives an indication of the stability of the sleep-wake rhythm across days, and varies from zero (low stability) to 1 (high stability). IS was derived by the ratio between the variance of the average 24-hour pattern around the mean and the overall variance. Higher values indicated stable rhythm. IS was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average last 7 nights of treatment was reported.
Time Frame: Baseline, Week 4
Population: FAS included group of randomized participants who received at least 1 dose of randomized study drug and had at least 1 postdose efficacy measurement. Participants who were evaluable for this measure at given time point were included for the assessment.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
ratio
  Baseline | 0.45 (0.173) | 0.47 (0.111) | 0.49 (0.118) | 0.46 (0.160) | 0.41 (0.104)
  Change at Week 4: number analyzed (Participants) | 7 | 10 | 8 | 8 | 9
  Change at Week 4 | 0.02 (0.098) | 0.01 (0.119) | 0.08 (0.092) | 0.03 (0.127) | 0.00 (0.102)
Statistical Analysis 1: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 2.5 mg; Test type: Superiority; p = 0.2991, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -0.032, 95% CI 2-sided [-0.094 to 0.029]
Statistical Analysis 2: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 5 mg; Test type: Superiority; p = 0.2861, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 0.033, 95% CI 2-sided [-0.028 to 0.095]
Statistical Analysis 3: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.0938, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -0.052, 95% CI 2-sided [-0.113 to 0.009]
Statistical Analysis 4: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 15 mg; Test type: Superiority; p = 0.8618, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 0.005, 95% CI 2-sided [-0.055 to 0.066]

33. Primary Outcome: Core Phase: Change From Baseline in Average Activity Counts Across Least Active 5-hour Period (L5) Per 24-Hour Period Over Week 1 of Treatment
Description: L5 was defined as the average activity across the least active 5-hour period per 24-hour period, with high values indicating restlessness. This value provides an indication of how restful (inactive) and regular the sleep periods are. L5 was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average first 7 nights of treatment was reported.
Time Frame: Baseline, Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: activity count
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
activity count
  Baseline | 1163.5 (373.3) | 1266.4 (678.1) | 1163.2 (591.8) | 1257.1 (836.6) | 1490.4 (963.1)
  Change at Week 1: number analyzed (Participants) | 12 | 11 | 13 | 11 | 12
  Change at Week 1 | 200.9 (633.3) | -259.8 (450.3) | -243.2 (333.6) | -211.6 (378.3) | -434.2 (509.1)

34. Primary Outcome: Core Phase: Change From Baseline in Average Activity Counts Across L5 Per 24-Hour Period Over Week 2 of Treatment
Description: L5 was defined as the average activity across the least active 5-hour period per 24-hour period, with high values indicating restlessness. This value provides an indication of how restful (inactive) and regular the sleep periods are. L5 was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average second 7 nights of treatment was reported.
Time Frame: Baseline, Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: activity count
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
activity count
  Baseline | 1163.5 (373.3) | 1266.4 (678.1) | 1163.2 (591.8) | 1257.1 (836.6) | 1490.4 (963.1)
  Change at Week 2: number analyzed (Participants) | 12 | 9 | 12 | 12 | 11
  Change at Week 2 | 85.8 (525.3) | -259.8 (244.9) | -218.7 (321.6) | 218.5 (455.9) | -246.1 (637.6)

35. Primary Outcome: Core Phase: Change From Baseline in Average Activity Counts Across L5 Per 24-Hour Period Over Week 3 of Treatment
Description: L5 was defined as the average activity across the least active 5-hour period per 24-hour period, with high values indicating restlessness. This value provides an indication of how restful (inactive) and regular the sleep periods are. L5 was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average third 7 nights of treatment was reported.
Time Frame: Baseline, Week 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: activity count
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
activity count
  Baseline | 1163.5 (373.3) | 1266.4 (678.1) | 1163.2 (591.8) | 1257.1 (836.6) | 1490.4 (963.1)
  Change at Week 3: number analyzed (Participants) | 11 | 11 | 12 | 12 | 12
  Change at Week 3 | 299.2 (1070.2) | -265.3 (507.0) | -233.0 (369.3) | -114.6 (376.6) | -396.1 (543.9)

36. Primary Outcome: Core Phase: Change From Baseline in Average Activity Counts Across L5 Per 24-Hour Period Over Week 4 of Treatment
Description: L5 was defined as the average activity across the least active 5-hour period per 24-hour period, with high values indicating restlessness. This value provides an indication of how restful (inactive) and regular the sleep periods are. L5 was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average last 7 nights of treatment was reported.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: activity count
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
activity count
  Baseline | 1163.5 (373.3) | 1266.4 (678.1) | 1163.2 (591.8) | 1257.1 (836.6) | 1490.4 (963.1)
  Change at Week 4: number analyzed (Participants) | 7 | 10 | 8 | 8 | 9
  Change at Week 4 | 293.1 (662.6) | -334.0 (476.4) | -344.5 (419.1) | 30.5 (772.5) | -160.7 (471.3)
Statistical Analysis 1: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 2.5 mg; Test type: Superiority; p = 0.0294, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -389.873, 95% CI 2-sided [-739.177 to -40.569]
Statistical Analysis 2: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 5 mg; Test type: Superiority; p = 0.0243, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -402.994, 95% CI 2-sided [-751.670 to -54.319]
Statistical Analysis 3: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.4209, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -141.026, 95% CI 2-sided [-489.805 to 207.752]
Statistical Analysis 4: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 15 mg; Test type: Superiority; p = 0.0398, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -367.845, 95% CI 2-sided [-717.870 to -17.820]

37. Primary Outcome: Core Phase: Change From Baseline in the Average Activity Count During the Most Active 10-hour Period (M10) Per 24-Hour Period Over Week 1 of Treatment
Description: M10 was defined as the average activity during the most active 10-hour period per 24-hour period with low levels indicating inactivity. M10 was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average first 7 nights of treatment was reported.
Time Frame: Baseline, Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: activity count
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
activity count
  Baseline | 8560.4 (2631.2) | 11567.0 (4266.3) | 12158.1 (3639.9) | 10662.1 (5023.6) | 11460.5 (4954.3)
  Change at Week 1: number analyzed (Participants) | 12 | 12 | 13 | 11 | 12
  Change at Week 1 | 59.7 (1832.6) | -731.4 (3373.5) | 42.5 (1789.3) | -334.6 (2659.2) | -111.2 (2558.0)

38. Primary Outcome: Core Phase: Change From Baseline in the Average Activity Count During the M10 Per 24-Hour Period Over Week 2 of Treatment
Description: M10 was defined as the average activity during the most active 10-hour period per 24-hour period with low levels indicating inactivity. M10 was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average second 7 nights of treatment was reported.
Time Frame: Baseline, Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: activity count
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
activity count
  Baseline | 8560.4 (2631.2) | 11567.0 (4266.3) | 12158.1 (3639.9) | 10662.1 (5023.6) | 11460.5 (4954.3)
  Change at Week 2: number analyzed (Participants) | 12 | 9 | 12 | 12 | 11
  Change at Week 2 | 232.7 (1829.1) | -968.8 (2885.6) | -121.1 (2137.3) | -564.2 (1975.7) | -325.4 (1585.4)

39. Primary Outcome: Core Phase: Change From Baseline in the Average Activity Count During the M10 Per 24-Hour Period Over Week 3 of Treatment
Description: M10 was defined as the average activity during the most active 10-hour period per 24-hour period with low levels indicating inactivity. M10 was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average third 7 nights of treatment was reported.
Time Frame: Baseline, Week 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: activity count
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
activity count
  Baseline | 8560.4 (2631.2) | 11567.0 (4266.3) | 12158.1 (3639.9) | 10662.1 (5023.6) | 11460.5 (4954.3)
  Change at Week 3: number analyzed (Participants) | 11 | 11 | 12 | 12 | 12
  Change at Week 3 | 300.3 (2094.9) | -986.2 (3502.0) | 572.6 (2216.0) | -828.3 (1970.2) | -635.8 (2413.6)

40. Primary Outcome: Core Phase: Change From Baseline in the Average Activity Count During the M10 Per 24-Hour Period Over Week 4 of Treatment
Description: M10 was defined as the average activity during the most active 10-hour period per 24-hour period with low levels indicating inactivity. M10 was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average last 7 nights of treatment was reported.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: activity count
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
activity count
  Baseline | 8560.4 (2631.2) | 11567.0 (4266.3) | 12158.1 (3639.9) | 10662.1 (5023.6) | 11460.5 (4954.3)
  Change at Week 4: number analyzed (Participants) | 7 | 10 | 8 | 8 | 9
  Change at Week 4 | 1650.4 (1815.3) | -1392.1 (2249.3) | -477.4 (963.2) | 279.8 (2204.0) | -457.8 (1788.7)
Statistical Analysis 1: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 2.5 mg; Test type: Superiority; p = 0.1162, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -1276.180, 95% CI 2-sided [-2878.587 to 326.226]
Statistical Analysis 2: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 5 mg; Test type: Superiority; p = 0.7781, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 227.464, 95% CI 2-sided [-1382.850 to 1837.777]
Statistical Analysis 3: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.4255, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -620.581, 95% CI 2-sided [-2170.342 to 929.179]
Statistical Analysis 4: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 15 mg; Test type: Superiority; p = 0.4672, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -577.820, 95% CI 2-sided [-2160.337 to 1004.697]

41. Primary Outcome: Core Phase: Change From Baseline in Amplitude of the Rest-activity Rhythm (AMP) Over Week 1 of Treatment
Description: AMP was amplitude of rest-activity rhythm calculated as the difference between M10 and L5. L5 was defined as the average activity across the least active 5-hour period per 24-hour period, with high values indicating restlessness. M10 was defined as the average activity during the most active 10-hour period per 24-hour period with low levels indicating inactivity. AMP was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average first 7 nights of treatment was reported.
Time Frame: Baseline, Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: activity count
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
activity count
  Baseline | 7396.9 (2728.3) | 10300.6 (4235.8) | 10994.8 (3601.8) | 9405.0 (5133.9) | 9970.0 (4905.8)
  Change at Week 1: number analyzed (Participants) | 12 | 11 | 13 | 11 | 12
  Change at Week 1 | -141.1 (1583.8) | -471.6 (3414.4) | 285.8 (1788.6) | -123.0 (2784.1) | 323.0 (2436.0)

42. Primary Outcome: Core Phase: Change From Baseline in AMP Over Week 2 of Treatment
Description: AMP was amplitude of rest-activity rhythm calculated as the difference between M10 and L5. L5 was defined as the average activity across the least active 5-hour period per 24-hour period, with high values indicating restlessness. M10 was defined as the average activity during the most active 10-hour period per 24-hour period with low levels indicating inactivity. AMP was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average second 7 nights of treatment was reported.
Time Frame: Baseline, Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: activity count
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
activity count
  Baseline | 7396.9 (2728.3) | 10300.6 (4235.8) | 10994.8 (3601.8) | 9405.0 (5133.9) | 9970.0 (4905.8)
  Change at Week 2: number analyzed (Participants) | 12 | 9 | 12 | 12 | 11
  Change at Week 2 | 146.8 (1603.7) | -708.9 (2934.6) | 97.6 (2105.2) | -782.7 (2141.4) | -79.3 (1672.5)

43. Primary Outcome: Core Phase: Change From Baseline in AMP Over Week 3 of Treatment
Description: AMP was amplitude of rest-activity rhythm calculated as the difference between M10 and L5. L5 was defined as the average activity across the least active 5-hour period per 24-hour period, with high values indicating restlessness. M10 was defined as the average activity during the most active 10-hour period per 24-hour period with low levels indicating inactivity. AMP was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average third 7 nights of treatment was reported.
Time Frame: Baseline, Week 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: activity count
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
activity count
  Baseline | 7396.9 (2728.3) | 10300.6 (4235.8) | 10994.8 (3601.8) | 9405.0 (5133.9) | 9970.0 (4905.8)
  Change at Week 3: number analyzed (Participants) | 11 | 11 | 12 | 12 | 12
  Change at Week 3 | 1.1 (1862.7) | -721.0 (3502.2) | 805.6 (2195.6) | -713.7 (2178.3) | -239.7 (2592.5)

44. Primary Outcome: Core Phase: Change From Baseline in AMP Over Week 4 of Treatment
Description: AMP was amplitude of rest-activity rhythm calculated as the difference between M10 and L5. L5 was defined as the average activity across the least active 5-hour period per 24-hour period, with high values indicating restlessness. M10 was defined as the average activity during the most active 10-hour period per 24-hour period with low levels indicating inactivity. AMP was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average last 7 nights of treatment was reported.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: activity count
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
activity count
  Baseline | 7396.9 (2728.3) | 10300.6 (4235.8) | 10994.8 (3601.8) | 9405.0 (5133.9) | 9970.0 (4905.8)
  Change at Week 4: number analyzed (Participants) | 7 | 10 | 8 | 8 | 9
  Change at Week 4 | 1357.3 (1801.9) | -1058.0 (2170.9) | -132.9 (840.7) | 249.4 (2694.7) | -297.1 (1608.2)
Statistical Analysis 1: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 2.5 mg; Test type: Superiority; p = 0.2984, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -839.088, 95% CI 2-sided [-2440.854 to 762.678]
Statistical Analysis 2: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 5 mg; Test type: Superiority; p = 0.4218, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 651.922, 95% CI 2-sided [-962.835 to 2266.678]
Statistical Analysis 3: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.5655, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -447.245, 95% CI 2-sided [-1998.440 to 1103.950]
Statistical Analysis 4: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 15 mg; Test type: Superiority; p = 0.8686, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = -130.603, 95% CI 2-sided [-1706.478 to 1445.272]

45. Primary Outcome: Core Phase: Change From Baseline in Relative Amplitude in the Rest-activity Rhythm (RA) Over Week 1 of Treatment
Description: RA was relative amplitude of the rest-activity rhythm calculated as the difference between M10 and L5 divided by M10 plus L5. L5 was defined as the average activity across the least active 5-hour period per 24-hour period, with high values indicating restlessness. M10 was defined as the average activity during the most active 10-hour period per 24-hour period with low levels indicating inactivity. RA was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average first 7 nights of treatment was reported.
Time Frame: Baseline, Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
ratio
  Baseline | 0.73 (0.136) | 0.79 (0.141) | 0.82 (0.089) | 0.77 (0.165) | 0.76 (0.148)
  Change at Week 1: number analyzed (Participants) | 12 | 11 | 13 | 11 | 12
  Change at Week 1 | -0.02 (0.101) | 0.01 (0.080) | 0.03 (0.067) | 0.02 (0.096) | 0.07 (0.073)

46. Primary Outcome: Core Phase: Change From Baseline in RA Over Week 2 of Treatment
Description: RA was relative amplitude of the rest-activity rhythm calculated as the difference between M10 and L5 divided by M10 plus L5. L5 was defined as the average activity across the least active 5-hour period per 24-hour period, with high values indicating restlessness. M10 was defined as the average activity during the most active 10-hour period per 24-hour period with low levels indicating inactivity. RA was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average second 7 nights of treatment was reported.
Time Frame: Baseline, Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
ratio
  Baseline | 0.73 (0.136) | 0.79 (0.141) | 0.82 (0.089) | 0.77 (0.165) | 0.76 (0.148)
  Change at Week 2: number analyzed (Participants) | 12 | 9 | 12 | 12 | 11
  Change at Week 2 | -0.00 (0.073) | 0.01 (0.063) | 0.03 (0.052) | -0.05 (0.112) | 0.05 (0.091)

47. Primary Outcome: Core Phase: Change From Baseline in RA Over Week 3 of Treatment
Description: RA was relative amplitude of the rest-activity rhythm calculated as the difference between M10 and L5 divided by M10 plus L5. L5 was defined as the average activity across the least active 5-hour period per 24-hour period, with high values indicating restlessness. M10 was defined as the average activity during the most active 10-hour period per 24-hour period with low levels indicating inactivity. RA was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average third 7 nights of treatment was reported.
Time Frame: Baseline, Week 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
ratio
  Baseline | 0.73 (0.136) | 0.79 (0.141) | 0.82 (0.089) | 0.77 (0.165) | 0.76 (0.148)
  Change at Week 3: number analyzed (Participants) | 11 | 11 | 12 | 12 | 12
  Change at Week 3 | -0.01 (0.143) | 0.01 (0.088) | 0.04 (0.063) | 0.01 (0.090) | 0.06 (0.080)

48. Primary Outcome: Core Phase: Change From Baseline in RA Over Week 4 of Treatment
Description: RA was relative amplitude of the rest-activity rhythm calculated as the difference between M10 and L5 divided by M10 plus L5. L5 was defined as the average activity across the least active 5-hour period per 24-hour period, with high values indicating restlessness. M10 was defined as the average activity during the most active 10-hour period per 24-hour period with low levels indicating inactivity. RA was determined by Actigraphy. Actigraphy was performed with an accelerometer that was worn on the wrist like a watch. It was programmed to monitor degree and intensity of movements while the device was being worn. Change from baseline to average last 7 nights of treatment was reported.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
ratio
  Baseline | 0.73 (0.136) | 0.79 (0.141) | 0.82 (0.089) | 0.77 (0.165) | 0.76 (0.148)
  Change at Week 4: number analyzed (Participants) | 7 | 10 | 8 | 8 | 9
  Change at Week 4 | -0.00 (0.117) | 0.01 (0.060) | 0.05 (0.049) | 0.01 (0.136) | 0.02 (0.069)
Statistical Analysis 1: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 2.5 mg; Test type: Superiority; p = 0.4638, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 0.020, 95% CI 2-sided [-0.034 to 0.074]
Statistical Analysis 2: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 5 mg; Test type: Superiority; p = 0.0322, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 0.060, 95% CI 2-sided [0.005 to 0.115]
Statistical Analysis 3: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.9144, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 0.003, 95% CI 2-sided [-0.051 to 0.056]
Statistical Analysis 4: Comparison: Core Phase: Lemborexant-matched Placebo vs Core Phase: Lemborexant 15 mg; Test type: Superiority; p = 0.0364, MMRM — Based on a MMRM analysis adjusted for baseline value, country, visit and treatment by visit interaction; LSM Difference = 0.057, 95% CI 2-sided [0.004 to 0.110]

49. Other Pre Specified Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: First dose of study drug (Day 1) to 14 days after last dose of study drug (approximately up to 2 years 7 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Extension Phase: Lemborexant 5 mg: Participants who completed the core study EOS visit within 30 days prior to enrollment in extension phase were eligible to participate in extension phase. Participants received one lemborexant 5 mg, tablet, orally, once daily, immediately (within 5 minutes) before the bedtime at night until lemborexant is commercially available, or until the lemborexant clinical development program for ISWRD is discontinued or up to 30 months.
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg | Extension Phase: Lemborexant 5 mg | Extension Phase: Lemborexant 10 mg | Extension Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12 | 5 | 14 | 6
Participants
  TEAEs | 4 | 3 | 3 | 4 | 6 | 4 | 10 | 5
  SAEs | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1

50. Other Pre Specified Outcome: Core Phase: Number of Participants in Each Category With Clinician's Global Impression of Change-Irregular Sleep-Wake Rhythm Disorder (CGIC-ISWRD) Global Score at Day 29
Description: The CGIC-ISWRD scale is a validated categorical measure of change in the participant's clinical condition between baseline and follow-up visits. It relies on both direct examination of the participant and an interview of the informant. The instrument consisted of 3 parts: a guided baseline interview administered to the participant and an informant, a follow-up interview administered to the participant and an informant, and a clinician's rating review. The baseline interview served as a reference for future ratings. During the baseline interview, the rater evaluated participant regarding domains of (1) sleep and wake symptoms; (2) mood and behavioral symptoms; (3) attention/arousal; and (4) social functioning. In the follow-up interview, a 7-pointscale was used, from 1 = marked improvement, 4 = no change, to 7 = marked worsening, to score each of the 4 domains and to provide a global score (1 [marked improvement] to 7 [marked worsening]).
Time Frame: Day 29
Population: The FAS included group of randomized participants who received at least 1 dose of randomized study drug and had at least 1 postdose efficacy measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
Participants
  Global score: Marked improvement | 1 | 0 | 0 | 0 | 0
  Global score: Moderate improvement | 1 | 0 | 2 | 1 | 0
  Global score: Minimal improvement | 4 | 4 | 4 | 5 | 3
  Global score: No change | 6 | 5 | 4 | 3 | 7
  Global score: Minimal worsening | 0 | 3 | 2 | 3 | 1
  Global score : Moderate worsening | 0 | 0 | 0 | 0 | 0
  Global score : Marked worsening | 0 | 0 | 0 | 0 | 0

51. Other Pre Specified Outcome: Core Phase: Change From Baseline in the Neuropsychiatric Inventory (NPI-10) Total Score at Day 29
Description: The NPI-10 assessed a wide range of behaviors seen in dementia for both frequency and severity. It is a 10 item questionnaire with the following domains: delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/liability and aberrant motor behavior. The total score was summarized and analyzed. This scale was administered with the caregiver as proxy for the participant. The total score was a sum of the 10 domains, where the score of each domain was calculated as frequency (scale: 1=occasionally to 4=very frequently) * Severity (scale: 1=Mild to 3=Severe). Each domain has a maximum score of 12 and all domains were equally weighted for total score, thus the range for the total score is 0 to 120 with 0 being completely healthy to 120 which is the worse score participant could get.
Time Frame: Baseline, Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 12
score on a scale
  Baseline: number analyzed (Participants) | 12 | 12 | 12 | 13 | 11
  Baseline | 3.8 (4.13) | 13.1 (17.77) | 7.7 (12.32) | 6.4 (10.27) | 5.5 (5.73)
  Change at Day 29: number analyzed (Participants) | 12 | 12 | 12 | 13 | 10
  Change at Day 29 | -2.8 (3.64) | -3.4 (9.23) | -0.3 (5.85) | -3.4 (8.95) | 3.8 (13.02)

52. Other Pre Specified Outcome: Core Phase: Change From Baseline in the Sleep Disorders Inventory (SDI) Score at Day 29
Description: The SDI is an expanded version of one item of the NPI. It described the frequency, severity, and caregiver burden of sleep-disturbed behaviors during a period prior to its administration. The SDI consists of the 7 sub questions relating to sleep from the NPI sleep disturbance item. Each of the sub questions is a separate question with frequency, severity, and caregiver distress rated by the caregiver with respect to the patient-participant for the 2 weeks prior to the visit. The SDI score is derived as the product of the average of the frequency ratings and the average of the severity ratings (range: 0-12 [worst]).
Time Frame: Baseline, Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 11
score on a scale
  Baseline: number analyzed (Participants) | 12 | 12 | 12 | 13 | 11
  Baseline | 0.79 (0.692) | 1.24 (1.576) | 0.74 (0.653) | 0.66 (0.748) | 1.44 (1.708)
  Change at Day 29: number analyzed (Participants) | 12 | 12 | 12 | 13 | 11
  Change at Day 29 | -0.48 (1.078) | -0.10 (0.616) | -0.33 (0.503) | -0.09 (0.574) | -0.49 (1.220)

53. Other Pre Specified Outcome: Extension Phase: Change From Baseline in SDI Total Score.
Description: as for outcome 52
Time Frame: Baseline, Day 133, 223, 313, 343, 373, 403, 493, 583, 673, and 763
Population: The safety analysis set included the group of extension phase participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment in extension phase. Here overall number analyzed "N" are the participants who were evaluable for the outcome measure. Number analyzed "n" are the participants who were evaluable for the outcome measure for given categories.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extension Phase: Lemborexant 5 mg | Extension Phase: Lemborexant 10 mg | Extension Phase: Lemborexant 15 mg
Number analyzed (Participants) | 5 | 12 | 6
score on a scale
  Baseline | 1.36 (1.948) | 0.74 (0.728) | 1.45 (2.331)
  Change at Day 133 (Visit 9): number analyzed (Participants) | 1 | 8 | 3
  Change at Day 133 (Visit 9) | 1.40 | -0.45 (0.600) | -0.63 (0.473)
  Change at Day 223 (Visit 12): number analyzed (Participants) | 0 | 6 | 3
  Change at Day 223 (Visit 12) |  | -0.60 (0.693) | 0.17 (0.306)
  Change at Day 313 (Visit 15): number analyzed (Participants) | 0 | 4 | 3
  Change at Day 313 (Visit 15) |  | -0.65 (0.574) | -0.17 (1.266)
  Change at Day 343 (Visit 16): number analyzed (Participants) | 1 | 2 | 2
  Change at Day 343 (Visit 16) | 0.60 | 0.55 (1.061) | 0.45 (0.919)
  Change at Day 373 (Visit 17): number analyzed (Participants) | 0 | 1 | 0
  Change at Day 373 (Visit 17) |  | -0.20 |
  Change at Day 403 (Visit 18): number analyzed (Participants) | 0 | 5 | 4
  Change at Day 403 (Visit 18) |  | -0.50 (0.539) | -0.55 (0.656)
  Change at Day 493 (Visit 19): number analyzed (Participants) | 0 | 3 | 1
  Change at Day 493 (Visit 19) |  | -0.13 (0.115) | -0.10
  Change at Day 583 (Visit 20): number analyzed (Participants) | 0 | 2 | 2
  Change at Day 583 (Visit 20) |  | -0.15 (0.071) | -0.35 (0.354)
  Change at Day 673 (Visit 21): number analyzed (Participants) | 0 | 1 | 2
  Change at Day 673 (Visit 21) |  | -0.30 | -0.15 (0.071)
  Change at Day 763 (Visit 22): number analyzed (Participants) | 0 | 2 | 0
  Change at Day 763 (Visit 22) |  | -0.05 (0.354) |

ADVERSE EVENTS:
Time Frame: First dose of study drug (Day 1) to 14 days after last dose of study drug (approximately up to 2 years 7 months)
Arm/Group | Core Phase: Lemborexant-matched Placebo | Core Phase: Lemborexant 2.5 mg | Core Phase: Lemborexant 5 mg | Core Phase: Lemborexant 10 mg | Core Phase: Lemborexant 15 mg | Extension Phase: Lemborexant 5 mg | Extension Phase: Lemborexant 10 mg | Extension Phase: Lemborexant 15 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/13 | 0/13 | 0/12 | 0/5 | 0/14 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/13 | 0/13 | 0/12 | 1/5 | 2/14 | 1/6
Other Adverse Events (participants affected / at risk) | 4/12 | 3/12 | 3/13 | 4/13 | 6/12 | 4/5 | 10/14 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Phase: Lemborexant-matched Placebo (N=12) | Core Phase: Lemborexant 2.5 mg (N=12) | Core Phase: Lemborexant 5 mg (N=13) | Core Phase: Lemborexant 10 mg (N=13) | Core Phase: Lemborexant 15 mg (N=12) | Extension Phase: Lemborexant 5 mg (N=5) | Extension Phase: Lemborexant 10 mg (N=14) | Extension Phase: Lemborexant 15 mg (N=6)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ilium fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Phase: Lemborexant-matched Placebo (N=12) | Core Phase: Lemborexant 2.5 mg (N=12) | Core Phase: Lemborexant 5 mg (N=13) | Core Phase: Lemborexant 10 mg (N=13) | Core Phase: Lemborexant 15 mg (N=12) | Extension Phase: Lemborexant 5 mg (N=5) | Extension Phase: Lemborexant 10 mg (N=14) | Extension Phase: Lemborexant 15 mg (N=6)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Sedation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Libido increased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Genital injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/57/NCT03001557/Prot_002.pdf
  • Statistical Analysis Plan: Core Phase (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/57/NCT03001557/SAP_003.pdf
  • Statistical Analysis Plan: Extension Phase (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT03001557/SAP_004.pdf